CLINICAL TRIAL: NCT02188979
Title: GlideScope Videolaryngoscopy and Pre-Operative Assessment of El-Ganzouri Risk Index for Tracheal Intubation in Morbidly Obese Patients The Prospective Observational GLOBE Study
Brief Title: GlideScope With EGRI Assessment in Obese Patients
Acronym: GLOBE
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Elena Cagnazzi, Medical Doctor Anesthesiologist, Università degli Studi di Brescia
Other Study IDs: GLOBE
Record Dates: First submitted 2014-07-06; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Morbid Obesity
Keywords: airway; equipment - laryngoscopes; intubation - tracheal; obesity.
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
BACKGROUND Unpredicted difficult tracheal intubation (DTI) with Macintosh laryngoscopy occurs frequently in obese patients. We investigated the incidence of DTI using the GlideScope® videolaryngoscope (GVL) with an algorithm based on a pre-operative assessment with the El Ganzouri Risk Index (EGRI).

METHODS We prospectively enrolled morbidly obese patients (BMI>40 kg/m2) undergoing abdominal surgery. Patients were scheduled for flexible fibre optic bronchoscopic intubation (FFBI) or GVL intubation if the EGRI score was ≥7 or <7, respectively. The primary outcome was the occurrence of DTI that was defined as Cormack and Lehane (C&L) grades ≥III, Intubation Difficulty Scale (IDS)>5 and modified IDS (mIDS)>5. A numeric rating scale (NRS) was also used. Secondary outcomes included intubation success during the first attempt, the time to Cormack (TTC), the time to intubation (TTI), failure to intubate, oxygen desaturation and difficult ventilation.

DETAILED DESCRIPTION:
The EGRI, a multivariate risk index that combines seven variables associated with DTI, was evaluated in all patients during the pre-anaesthesia visit. The results were reported in the clinical chart. All tracheal intubations in obese patients needing surgery were routinely performed using GVL. The intubations were performed or assisted by five board-certified anaesthesiologists who had prior experience with at least 20 GVL intubations, as well as at least two years of experience with anaesthesia in obese patients. In cases where the GVL intubation was performed by anaesthesiologists that were in training, the GVL expert was actively advising the operator during all of the intubating procedures. The standard equipment included a GVL with blade number three to five and an orotracheal hockey stick tube with a malleable single-use stylet (Fr 14, Intubating Stylet, DEAS). The standard anaesthesia induction started with 3-5 minutes of pre-oxygenation using 5 cm H2O PEEP in a 30° head-up position, as well as induction with fentanyl 3 μg kg -1 (LBW), propofol 2-3 mg kg -1 (LBW) and suxamethonium 1 mg Kg -1 (TBW). When spontaneous respiration ceased, the patient was mask ventilated with 100% oxygen. The tube was lubricated and advanced into the mouth under direct visual guidance to avoid complications, and then, under indirect visual guidance using the GVL monitor. The correct placement of the cuffed tube was verified using a capnograph and a stethoscope. The tube sizes were 7.0 for women and 7.5 for men. Each patient was monitored using an electrocardiogram, non-invasive arterial blood pressure measurement, and pulse oximetry before both tracheal intubation and anaesthesia induction. The basic demographic data and airway characteristics necessary to evaluate the primary outcome and to calculate the EGRI score were registered prior to anaesthesia. Patients with an EGRI score of 7 or higher were scheduled for elective fibre optic flexible bronchoscopic intubation (FFBI), while patients with an EGRI score of less than 7 underwent anaesthesia induction and GVL intubation, according to a predefined algorithm

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI)>40 kg m-2.
* Surgery with tracheal intubation scheduled

Exclusion Criteria:

* age < 18 years
* severe psychological disorders that have the possibility of limiting the patient's comprehension of information
* previously impossible mask ventilation or intubation with GVL
* presence of pharyngo-laryngeal or neck tumours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our patients population is the population of morbidly obese patients scheduled for bariatric surgery or other non-bariatric abdominal surgical interventions and referring to the University Division of Anaesthesia and Intensive Care at Spedali Civili of Brescia.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of DTI that was defined as Cormack and Lehane (C&L) grades ≥III, Intubation Difficulty Scale (IDS)>5 and modified IDS (mIDS)>5. A numeric rating scale (NRS) was also used. | Ten minutes after the intubation
  The primary outcome was the incidence of DTI. Because scores specifically designed to assess DTI with GVL are not available, we used the Cormack and Lehane (C&L) grades ≥III, the Intubation Difficulty Scale (IDS) >5 and a modified IDS (mIDS) >5 to assess DTI. We also conducted a subjective assessment of DTI as rated by the operator on a numeric rating scale (NRS), from 0 (easiest) to 10 (the most difficult procedure).

SECONDARY OUTCOMES:
frequency of tracheal intubation success during the first attempt | Ten minutes after the intubation
  The frequency of intubation success at the first attempt was defined as being when the tracheal intubation was successfully achieved with all the following criteria fulfilled: a single introduction of the laryngoscope and tube progression, C&L I or IIa without external laryngeal displacement, and no need for help by another operator.
the time to Cormack (TTC) and the time to tracheal intubation (TTI). | Ten minutes after the intubation
  TTC was measured from the time the instrument entered patient's mouth until the optimal laryngeal view. TTI was measured from the time the instrument entered the patient's mouth until the tube cuff inflation.
intubation failures | Ten minutes after the intubation failure
  Failure to intubate was defined as when tracheal intubation proved impossible after three attempts
difficult mask ventilation | Ten minutes after the intubation
  Difficult ventilation was defined with the use of the Han scale
oxygen desaturation | Ten minutes after the intubation
  Oxygen desaturation was defined as an oxygen saturation of less than 90%

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Mosca, MD, Principal Investigator — Università degli Studi di Brescia; Elena Cagnazzi, MD, Principal Investigator — Università degli Studi di Brescia; Federico Pe, MD, Principal Investigator — Università degli Studi di Brescia; Tiziana Togazzari, MD, Study Chair — Universitry of Brescia; Ottavia Manenti, MD, Study Chair — Univertsity of Brescia; Francesco Mittempergher, MD, Study Chair — Università degli Studi di Brescia; Elena Raffetti, MD, Study Chair — Università degli Studi di Brescia; Francesco Donato, Professor, Study Chair — Università degli Studi di Brescia; Nicola Latronico, Professor, Study Director — Università degli Studi di Brescia
Locations (1):
- Department of Anaesthesia, Critical Care Medicine and Emergency University of Brescia at Spedali Civili., Brescia, Brescia, Italy

REFERENCES:
- [Background] Padwal RS, Klarenbach SW, Wang X, Sharma AM, Karmali S, Birch DW, Majumdar SR. A simple prediction rule for all-cause mortality in a cohort eligible for bariatric surgery. JAMA Surg. 2013 Dec;148(12):1109-15. doi: 10.1001/jamasurg.2013.3953. PMID 24132685
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery Worldwide 2008. Obes Surg. 2009 Dec;19(12):1605-11. doi: 10.1007/s11695-009-0014-5. PMID 19885707
- [Background] Nicholson A, Smith AF, Lewis SR, Cook TM. Tracheal intubation with a flexible intubation scope versus other intubation techniques for obese patients requiring general anaesthesia. Cochrane Database Syst Rev. 2014 Jan 17;2014(1):CD010320. doi: 10.1002/14651858.CD010320.pub2. PMID 24443105
- [Background] Cook TM, MacDougall-Davis SR. Complications and failure of airway management. Br J Anaesth. 2012 Dec;109 Suppl 1:i68-i85. doi: 10.1093/bja/aes393. PMID 23242753
- [Background] Juvin P, Lavaut E, Dupont H, Lefevre P, Demetriou M, Dumoulin JL, Desmonts JM. Difficult tracheal intubation is more common in obese than in lean patients. Anesth Analg. 2003 Aug;97(2):595-600. doi: 10.1213/01.ANE.0000072547.75928.B0. PMID 12873960
- [Background] Kim WH, Ahn HJ, Lee CJ, Shin BS, Ko JS, Choi SJ, Ryu SA. Neck circumference to thyromental distance ratio: a new predictor of difficult intubation in obese patients. Br J Anaesth. 2011 May;106(5):743-8. doi: 10.1093/bja/aer024. Epub 2011 Feb 24. PMID 21354999
- [Background] Serocki G, Neumann T, Scharf E, Dorges V, Cavus E. Indirect videolaryngoscopy with C-MAC D-Blade and GlideScope: a randomized, controlled comparison in patients with suspected difficult airways. Minerva Anestesiol. 2013 Feb;79(2):121-9. Epub 2012 Oct 2. PMID 23032922
- [Background] Cortellazzi P, Minati L, Falcone C, Lamperti M, Caldiroli D. Predictive value of the El-Ganzouri multivariate risk index for difficult tracheal intubation: a comparison of Glidescope videolaryngoscopy and conventional Macintosh laryngoscopy. Br J Anaesth. 2007 Dec;99(6):906-11. doi: 10.1093/bja/aem297. Epub 2007 Oct 25. PMID 17962241
- [Background] el-Ganzouri AR, McCarthy RJ, Tuman KJ, Tanck EN, Ivankovich AD. Preoperative airway assessment: predictive value of a multivariate risk index. Anesth Analg. 1996 Jun;82(6):1197-204. doi: 10.1097/00000539-199606000-00017. PMID 8638791
- [Background] Caldiroli D, Cortellazzi P. A new difficult airway management algorithm based upon the El Ganzouri Risk Index and GlideScope(R) videolaryngoscope. A new look for intubation? Minerva Anestesiol. 2011 Oct;77(10):1011-7. Epub 2011 May 24. PMID 21610665
- [Background] Cooper RM, Pacey JA, Bishop MJ, McCluskey SA. Early clinical experience with a new videolaryngoscope (GlideScope) in 728 patients. Can J Anaesth. 2005 Feb;52(2):191-8. doi: 10.1007/BF03027728. PMID 15684262
- [Background] Maassen R, Lee R, Hermans B, Marcus M, van Zundert A. A comparison of three videolaryngoscopes: the Macintosh laryngoscope blade reduces, but does not replace, routine stylet use for intubation in morbidly obese patients. Anesth Analg. 2009 Nov;109(5):1560-5. doi: 10.1213/ANE.0b013e3181b7303a. Epub 2009 Aug 27. PMID 19713258
- [Background] Serocki G, Bein B, Scholz J, Dorges V. Management of the predicted difficult airway: a comparison of conventional blade laryngoscopy with video-assisted blade laryngoscopy and the GlideScope. Eur J Anaesthesiol. 2010 Jan;27(1):24-30. doi: 10.1097/EJA.0b013e32832d328d. PMID 19809328
- [Background] Andersen LH, Rovsing L, Olsen KS. GlideScope videolaryngoscope vs. Macintosh direct laryngoscope for intubation of morbidly obese patients: a randomized trial. Acta Anaesthesiol Scand. 2011 Oct;55(9):1090-7. doi: 10.1111/j.1399-6576.2011.02498.x. Epub 2011 Sep 8. PMID 22092206
- [Background] Xue FS, Li CW, Zhang GH, Li XY, Sun HT, Liu KP, Liu J, Wang X. GlideScope-assisted awake fibreoptic intubation: initial experience in 13 patients. Anaesthesia. 2006 Oct;61(10):1014-5. doi: 10.1111/j.1365-2044.2006.04809.x. No abstract available. PMID 16978330
- [Background] Ydemann M, Rovsing L, Lindekaer AL, Olsen KS. Intubation of the morbidly obese patient: GlideScope((R)) vs. Fastrach. Acta Anaesthesiol Scand. 2012 Jul;56(6):755-61. doi: 10.1111/j.1399-6576.2012.02693.x. Epub 2012 Apr 23. PMID 22524487
- [Background] DeMaria EJ. Bariatric surgery for morbid obesity. N Engl J Med. 2007 May 24;356(21):2176-83. doi: 10.1056/NEJMct067019. No abstract available. PMID 17522401
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Adnet F, Borron SW, Racine SX, Clemessy JL, Fournier JL, Plaisance P, Lapandry C. The intubation difficulty scale (IDS): proposal and evaluation of a new score characterizing the complexity of endotracheal intubation. Anesthesiology. 1997 Dec;87(6):1290-7. doi: 10.1097/00000542-199712000-00005. PMID 9416711
- [Background] Han R, Tremper KK, Kheterpal S, O'Reilly M. Grading scale for mask ventilation. Anesthesiology. 2004 Jul;101(1):267. doi: 10.1097/00000542-200407000-00059. No abstract available. PMID 15220820
- [Background] Sun DA, Warriner CB, Parsons DG, Klein R, Umedaly HS, Moult M. The GlideScope Video Laryngoscope: randomized clinical trial in 200 patients. Br J Anaesth. 2005 Mar;94(3):381-4. doi: 10.1093/bja/aei041. Epub 2004 Nov 26. PMID 15567809
- [Background] Aziz MF, Healy D, Kheterpal S, Fu RF, Dillman D, Brambrink AM. Routine clinical practice effectiveness of the Glidescope in difficult airway management: an analysis of 2,004 Glidescope intubations, complications, and failures from two institutions. Anesthesiology. 2011 Jan;114(1):34-41. doi: 10.1097/ALN.0b013e3182023eb7. PMID 21150569
- [Background] Caldiroli D, Molteni F, Sommariva A, Frittoli S, Guanziroli E, Cortellazzi P, Orena EF. Upper limb muscular activity and perceived workload during laryngoscopy: comparison of Glidescope(R) and Macintosh laryngoscopy in manikin: an observational study. Br J Anaesth. 2014 Mar;112(3):563-9. doi: 10.1093/bja/aet347. Epub 2013 Oct 22. PMID 24148322